CLINICAL TRIAL: NCT06126679
Title: Effectiveness and Cost Effectiveness of a 1-year Dietary and Physical Activity Intervention of Childhood Obesity - Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Hyvinkää Childhood Obesity Study (HCOS), Randomized Controlled Clinical Trial for Effectiveness and Costs of a 1-year Lifestyle Intervention.
Acronym: HCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anni Martikainen, clinical nutritionist, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASLI
Record Dates: First submitted 2023-10-09; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: 80 children are recruited for this study and they randomize either to an intervention group or a control group with standard care. Intervention group receive intensive, family-based diet and physical activity counseling, deliver by a multidisciplinary team of a pediatrician, a nurse and a clinical nutritionist. Control group do not receive any lifestyle intervention during the study. The inclusion criteria are weight-for-height ≥+40% or ≥+30% and increasing and age of 6-12 years. All participants fill out the study questionnaires and plasma samples are taken at baseline and at 12 months. Outcome variables will be compared between intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The 1-year lifestyle intervention includes intensive, family-based diet and physical activity counselling. The multidisciplinary team consists of one pediatrician, one specialist nurse and a clinical nutritionist. Children with their parents meet the pediatrician two times, the specialist nurse five times and the clinical nutritionist three times during the 1-year intervention. One of the meetings with the clinical nutritionist is only for parents and the child is with the nurse at the same time.
  The treatment is based on educational and behavioural counselling and motivating the participants to change their lifestyle and to support the parents in managing their children´s behaviour. The aim of counselling is to increase awareness of healthy dietary and physical activity habits; to achieve a suitable energy balance, to create a positive attitude to physical activity, to promote optimal sleep duration and to improve the children´s body image and body control.
  Interventions: Procedure: 1-year dietary and physical activity intervention of childhood obesity
- control group (No Intervention): Participants in the control group continue with the standard care in primary care and do not receive any special lifestyle intervention during the study.

INTERVENTIONS:
Procedure: 1-year dietary and physical activity intervention of childhood obesity — The 1-year lifestyle intervention includes intensive, family-based diet and physical activity counselling. Children with their parents meet the pediatrician two times, the specialist nurse five times and the clinical nutritionist three times during the 1-year intervention. One of the meetings with the clinical nutritionist is only for parents and the child is with the nurse at the same time.
  The participants in the intervention group are advised and motivated to increase their regular daily physical activity and to reduce sedentary habits. They have one group session for the training in the gymnasium with physical education instructor. The physical education instructor gives a voluntary lecture for parents about increasing physical activity and reducing sedentary time.
  Arms: intervention group

SUMMARY:
The aim of this study is to evaluate the effects of lifestyle intervention on the management of childhood overweight and to explore the factors that contribute to the outcome, as well as the costs for the health care system. The hypotheses of the study are that lifestyle intervention is efficient in reducing BMI-SDS and thus effective in preventing overweight to progress to obesity, and it is also cost effective.

The research is necessary for the development of overweight treatment, and try to find out the optimal duration and intensity for the treatment and content useful for clinical work.

DETAILED DESCRIPTION:
Methods and analyses: The aim of this study is to recruit 80 children and to randomize them either to an intervention group or a control group with standard care. Intervention group receive intensive, family-based diet and physical activity counseling, deliver by a multidisciplinary team of a pediatrician, a nurse and a clinical nutritionist. Control group do not receive any lifestyle intervention during the study. The inclusion criteria are weight-for-height ≥+40% or ≥+30% and increasing and age of 6-12 years. All participants fill out the study questionnaires and plasma samples are taken at baseline and at 12 months. Outcome variables will be compared between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

weight for height at least + 40 % or ≥ 30 % and it is rising

Exclusion Criteria:

Clinical diagnosis of endocrine or mental diseases.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the efficacy of the intervention for the ISO-BMI | 12 months
  How much ISO-BMI change during the intervention (kg/m2)
The costs of the intervention for the health care system | 12 months
  Investigators calculate the costs (euros) of the intervention (the price of research visits, laboratory tests, the salary of emplyees and the cost of research rooms).

CONTACTS AND LOCATIONS:
Overall Officials: Anni Martikainen, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Non-operative Services, Internal Medicine and Rehabilitation, Clinical Nutrition Hyvinkää Hospital, Hyvinkää, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martikainen A, Eloranta AM, Schwab U, Ormala T. Effectiveness and cost-effectiveness of a 1-year dietary and physical activity intervention of childhood obesity-study protocol for a randomized controlled clinical trial. Trials. 2024 Jul 27;25(1):508. doi: 10.1186/s13063-024-08348-7. PMID 39068465